CLINICAL TRIAL: NCT07101692
Title: The Effect of Virtual Reality in Teaching Nasogastric Catheter Application Skills to New Graduate Nurses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Eminoğlu (Other)
Responsible Party: Sponsor-Investigator, Ayşe Eminoğlu, Research Assistant, Gaziantep Islam Science and Technology University
Organization: Gaziantep Islam Science and Technology University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 28.07.2025-1; Gaziantep Islam Science and Te (Other: Gaziantep Islam Science and Tecnology)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Nurses
Keywords: nursing; virtual realtiy; nasogastric catheter

STUDY DESIGN:
Intervention Model Description: This research will be conducted in two stages: design and implementation. In the first stage of the research, nasogastric catheter application skill reminder training, preparation of knowledge test, skill checklist and measurement tools, realization of software suitable for virtual reality glasses according to nasogastric catheter application process steps and integration into the glasses are included. In the second phase of the study, it is planned to evaluate the knowledge, skills, self-confidence, anxiety and motivation of the control and experimental groups with the intervention applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental Group (Experimental): - The experimental group will perform the nasogastric catheter insertion skill with 3D virtual reality glasses.
  Interventions: Behavioral: Virtual Reality-Based NGT Training
- Behavioral: virtual reality (Experimental): - The control group will try the nasogastric catheter insertion skill 3 times on their own.
  Interventions: Behavioral: Virtual Reality-Based NGT Training

INTERVENTIONS:
Behavioral: Virtual Reality-Based NGT Training — Participants will be given nasogastric catheter application training accompanied by a PowerPoint presentation and then they will be provided with three individual applications on the model.

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effectiveness of virtual reality (VR) technology in teaching nasogastric catheter (NGS) application skills to newly graduated nurses. The study will be conducted with nurses working at Eskişehir Osmangazi University Health Practice and Research Hospital. Participants will be divided into experimental (VR-assisted training) and control (traditional training) groups through randomization. After the training, knowledge level, skill score, self-confidence, anxiety and motivation levels of both groups will be compared. Data collection tools include knowledge test, skills checklist and visual comparison scales. The study aims to reveal the effects of integration of virtual reality technology into nursing education on clinical skill development.

DETAILED DESCRIPTION:
Health services play a critical role in improving the quality of life of people and nurses play an important role in the provision of these services. Nursing is a profession that requires a high level of practical competence as well as clinical knowledge and skills (Polat, 2024). The ability of nurses to provide effective patient care is directly related to the effectiveness of their education processes. Providing education processes with high quality and modern methods is critical for nurses to improve their clinical skills and reinforce their professional identities (Kara, 2024). Nasogastric catheter (NGS) application, which is one of these skills, is an important practice in meeting the nutritional needs of patients in many clinical situations. Nurses need to apply this skill correctly and safely in order for patients to be fed properly and the treatment process to function properly (Şendir & Kızıl, 2019). However, learning NGS application skills requires practical experience as well as theoretical knowledge. Especially newly graduated nurses may face various difficulties in developing such clinical skills. Inadequate educational environments, low number of cases and limited opportunities for practicing lead to difficulties for newly graduated nurses to acquire these skills. This situation may affect the professional competencies of nurses as well as the quality of patient care (Aygin & Yılmaz, 2022; Güngör et al., 2023; Kulakaç & Çilingir, 2023).

In addition to traditional training methods, virtual reality (VR) technology stands out as a revolutionary tool in teaching clinical skills. Virtual reality allows nurses to make mistakes and improve their skills in a safe environment before experiencing risky practices in the real world. VR can support nurses to learn clinical skills more effectively, practice and make the right decisions. In this context, virtual reality-based training materials can be used to gain NGS application skills (Sarıkoç, 2016).However, research to determine the impact of virtual reality on nursing is still limited. A more in-depth examination of how virtual reality is used in nursing, its effects on nurses, and the potential benefits of this technology on the teaching of clinical skills will make a significant contribution to the nursing profession. In particular, investigating the effectiveness of virtual reality technology for new graduate nurses to improve their nasogastric catheterization skills may improve the use of technology in nursing education and increase the safety of pre-nurses in clinical skills (Chang et al., 2024).

This study aims to determine the role of virtual reality in education, emphasize the benefits of this technology in clinical skills training, and provide suggestions to increase student success in the education process. In addition, a comparison of traditional training methods and virtual reality-based training methods will reveal the advantages and limitations of both approaches. This research will provide a valuable resource to modernize educational processes and enable nurses to develop their clinical skills more efficiently by providing a new perspective on skill performance in nursing. In this context, the aim of the study was to investigate the effectiveness of teaching nasogastric catheterization skills of new graduate nurses with virtual reality technology.

ELIGIBILITY:
Inclusion Criteria:

* Working in internal and surgical clinics,
* Volunteering to participate in the research,
* Over 18 years of age.

Exclusion Criteria:

* Working in outpatient clinics, physical therapy, psychiatry and pediatric clinics,
* Participate in group work,
* The nurse volunteered to participate in the study and then wanted to withdraw from the study,
* Filling the data collection forms of the research incompletely,
* Having any disability that would prevent answering the survey questions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nasogastric Catheter Application Skill Score | 7 day
  The change in the mean score of the nasogastric catheter application skill checklist (pre-test and post-test comparison) will be evaluated with the application on the model in the first week after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Eminoğlu, Dr., Study Director — ayse.eminoglu@gibtu.edu.tr
Locations (1):
- Gaziantep Islam Science and Technology, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not planned to share the individual participant data (IPD) collected in this study with other researchers. IPD will not be shared in accordance with the principles of participant privacy protection and data security.